CLINICAL TRIAL: NCT07273214
Title: Knowledge, Attitude and Practice of Third Trimester Pregnant Mothers Towards Self-Medication in Assiut, Egypt: A Cross-Sectional Observational Study
Brief Title: Knowledge, Attitude and Practice of Third Trimester Pregnant Mothers Towards Self-Medication in Assiut, Egypt
Acronym: SM-PREG
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, May Mohamed Abdelwahab Mohmoud, Resident, Obstetric and Gynecology Department, Assiut University
Other Study IDs: SM-PREG-ASSIUT-2025
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Third Trimeser
Keywords: anaemia; pregnancy; diabetis
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Third-trimester pregnant women (Assiut ANC cohort): A single observational cohort of pregnant women in their third trimester (≥ 28 weeks gestation) who attend antenatal care (ANC) clinics at Assiut University Hospital and selected primary health centers in Assiut, Egypt. Participants are interviewed once using a structured, pretested, interviewer-administered questionnaire to assess knowledge, attitude and practice (KAP) regarding self-medication during pregnancy, types of medicines used, reasons for use, and sources of information. Data collection is non-interventional and confidentiality is maintained.
  Interventions: Other: Structured Questionnaire on Self-Medication During Pregnancy

INTERVENTIONS:
Other: Structured Questionnaire on Self-Medication During Pregnancy — A structured, pretested interviewer-administered questionnaire designed to assess the knowledge, attitude, and practice (KAP) of pregnant women in their third trimester regarding self-medication during pregnancy. The tool includes sections on sociodemographic data, pregnancy history, knowledge of medication use, attitudes toward drug safety, and patterns of self-medication. It is used once during a single face-to-face interview. No drug, biological, or device is administered.

SUMMARY:
This study aims to assess the knowledge, attitude, and practice (KAP) of third-trimester pregnant women toward self-medication in Assiut, Egypt. Self-medication is a common behavior among pregnant women, often influenced by cultural habits, easy access to medications, and limited awareness of potential risks.

Through a structured, interviewer-administered questionnaire, this cross-sectional study will collect data on the prevalence and pattern of self-medication, types of medications used, reasons for use, and sources of information. Participants will be recruited from antenatal care (ANC) clinics at Assiut University Hospital and selected primary health care centers.

The findings of this research will help identify gaps in awareness and guide educational interventions to promote safe medication practices during pregnancy.

DETAILED DESCRIPTION:
Self-medication during pregnancy is a significant public health concern, as inappropriate use of medications can lead to adverse maternal and fetal outcomes. In developing countries, including Egypt, the availability of over-the-counter drugs, social beliefs, and lack of regulatory control contribute to this problem. However, data describing the magnitude and determinants of self-medication among pregnant women in Upper Egypt are limited.

This prospective cross-sectional study will be conducted among third-trimester pregnant women attending antenatal clinics at Assiut University Hospital and selected primary health care centers in Assiut, Egypt. A structured, pretested questionnaire will be used to collect data through face-to-face interviews by trained researchers.

The questionnaire covers sociodemographic data, obstetric history, knowledge about medication use during pregnancy, attitudes toward self-medication, and actual self-medication practices. It also includes items about commonly used drug types, sources of information, and reasons for self-medication.

A total of approximately 420 participants will be recruited using convenience sampling. Data will be analyzed using IBM SPSS version 29. Descriptive and inferential statistics will be applied to identify significant associations between self-medication practices and participant characteristics.

The study aims to:

Determine the prevalence of self-medication among third-trimester pregnant women.

Assess knowledge and attitudes regarding medication safety during pregnancy.

Identify the common drugs used and reasons for self-medication.

Provide recommendations for awareness and health education programs targeting pregnant women.

Ethical approval has been obtained from the Faculty of Medicine, Assiut University. Written informed consent will be obtained from all participants before enrollment. No intervention or experimental drug will be administered, and participant confidentiality will be maintained throughout the study.

The results of this research will contribute to improving antenatal care and maternal health policies by emphasizing the need for education about rational medication use during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the third trimester (≥28 weeks of gestation)
* Attending antenatal care at Assiut University Hospital or selected primary health centers during the study period
* Willing to participate and able to provide informed consent

Exclusion Criteria:

* Pregnant women with known psychiatric disorders or cognitive impairment that may affect questionnaire reliability.
* Women with severe obstetric complications requiring emergency management.
* Women unwilling to participate or unable to complete the interview.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The study population includes third-trimester pregnant women attending the antenatal care outpatient clinics at Assiut University Hospital and selected primary health care centers in Assiut Governorate, Egypt, during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Prevalence of self-medication among third-trimester pregnant women | from 28-40 weeks of gestation
  The primary outcome will be the proportion (%) of third-trimester pregnant women who report self-medicating with any pharmaceutical or herbal product during their current pregnancy. Data will be collected using a structured interviewer-administered questionnaire assessing medication type, reason for use, and source of information. Prevalence will be calculated as the number of women reporting self-medication divided by the total number of surveyed participants.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kashif MML, El-Tahty SE: An assessment of the factors influencing the use of over-the-counter medication during the second trimester of pregnancy, Egypt. Int J Nurs Sci. 2018, 12:99-107.
- [Result] World Health Organization, (2000). Guidelines for the regulatory assessment of medicinal products for use in self-medication. https://apps.who.int/iris/handle/10665/ 66154
- [Result] Hughes CM, McElnay JC, Fleming GF. Benefits and risks of self medication. Drug Saf. 2001;24(14):1027-37. doi: 10.2165/00002018-200124140-00002. PMID 11735659